CLINICAL TRIAL: NCT05436002
Title: Treatment of Buccal Ginvigal Recessions With the Tunnel Technique in Conjunction With Cross-linked Hyaluronic Acid and Subepithelial Connective Tissue Graft. A Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Vanessa Rocha Rodrigues, Dra, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cross-linked hyaluronic acid
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Cross-linked Hyaluronic Acid
Keywords: cross-linked hyaluronic acid; tunnel technique; gingival recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Cross-linked Hyaluronic Acid (Active Comparator): Tunnel Technique in Conjunction With Cross-linked Hyaluronic Acid and Subepithelial Connective Tissue Graft.
  Interventions: Device: With Cross-linked Hyaluronic Acid
- Whitout Cross-linked Hyaluronic Acid (Placebo Comparator): Tunnel Technique in Conjunction With Subepithelial Connective Tissue Graft.
  Interventions: Device: With Cross-linked Hyaluronic Acid

INTERVENTIONS:
Device: With Cross-linked Hyaluronic Acid — Without Cross-linked Hyaluronic Acid

SUMMARY:
To evaluate the outcomes of buccal gengival recession type 1 (RT1) treated with the tunnel technique in conjunction with a cross-linked hyaluronic acid and subepithelial palatal connective tissue grafts.

DETAILED DESCRIPTION:
To evaluate the outcomes of buccal gengival recession type 1 (RT1) treated with the tunnel technique in conjunction with a cross-linked hyaluronic acid and subepithelial palatal connective tissue grafts.

To evaluate the esthetic outcome as perceived by periodontists, using the root coverage esthetic score (RES).

Test Group - Tunnel technique in conjunction with a cross-linked hyaluronic acid and subepithelial palatal connective tissue grafts.

Control Group - Tunnel technique and subepithelial palatal connective tissue grafts.

ELIGIBILITY:
Inclusion Criteria:

* None of the patients were smokers and all were systemically healthy without any signs of periodontal disease.
* Each patient had to display at least one ginvigal recession (RT1) of a depth of ≥ 2 mm.
* Patients exhibited an adequate level of oral hygiene evidenced by a full- mouth plaque score (FMPS) < 25%39 and full-mouth bleeding score (FMBS) < 25%.

Exclusion Criteria:

* Smokers
* Gingival recesstion RT 2 or RT 3 (Cairo 2011).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Gingival margin | 6 month after surgery
  Score 0: failure of root coverage (gingival margin apical or equal to the baseline recession); Score 3: partial root coverage; Score 6: complete root coverage with no detectable CEJ.
Marginal tissue contour | 6 month after surgery
  Score 0: irregular gingival margin (it does not follow CEJ); Score 1: proper marginal contour/scalloped gingival margin (following CEJ).
Soft tissue texture | 6 month after surgery
  Score 0: presence of scar formation and/or keloid-like appearance; Score 1: absence of scar or keloid formation.
Mucogingival junction | 6 month after surgery
  Score 0: MGJ not aligned with MGJ on adjacent teeth; Score 1: MGJ aligned with MGJ on adjacent teeth.
Gingival color | 6 month after surgery
  Score 0: color of tissue differs from gingival color on adjacent teeth; Score 1: normal color and integration with the adjacent soft tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Rodrigues, Dr, Principal Investigator — University of Lisbon

IPD SHARING:
Plan to Share IPD: No